CLINICAL TRIAL: NCT02230800
Title: Randomised Double-blind Placebo Controlled Phase II Trial of Tocovid SupraBio in Combination With Pentoxifylline (PTX) in Patients Suffering Long-term Adverse Effects of Radiotherapy for Pelvic Cancer
Brief Title: PPALM-Palm Oil and Pentoxifylline Against Late Morbidity
Acronym: PPALM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Malaysia Palm Oil Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCR3894
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2019-12-23 (Actual); Status verified 2019-01

CONDITIONS: Long-term Adverse Effects of Radiotherapy for Pelvic Cancer
MeSH Terms: interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tocovid SupraBio plus pentoxifylline (PTX) (Experimental): Tocovid SupraBio* 200mg po bd plus pentoxifylline (PTX) 400mg po bd for 12 months.
  Interventions: Drug: Tocovid SupraBio plus pentoxifylline
- Matching placebos (Placebo Comparator): Matching placebos bd for 12 months.
  Interventions: Drug: Matching placebos

INTERVENTIONS:
Drug: Tocovid SupraBio plus pentoxifylline
  Arms: Tocovid SupraBio plus pentoxifylline (PTX)
Drug: Matching placebos
  Arms: Matching placebos

SUMMARY:
Side effects are common after treatment with radiotherapy for tumours in the pelvis and can affect the way the bowel and urinary system work as well as causing sexual difficulties, skin damage and bone problems. Problems in the bowel, bladder, sexual organs and skin mostly result from thickening of the tissues in response to radiotherapy, a process called "fibrosis". Fibrosis often worsens over time.

There has been progress in treating bowel symptoms which usually are the worst problem after radiotherapy. However, even after receiving the best possible treatments, while many patients are better, they are often not cured of all their difficult problems.

For some years, it has been hypothesised that if fibrosis could be treated then symptoms would improve. Recent research in laboratory animals has suggested that an effective treatment for radiation-induced fibrosis is combination therapy with a drug called Pentoxifylline together with a nutritional supplement containing gamma-tocotrienol (Tocovid SupraBio), a substance derived from palm oil. Both of these agents are simple to take and side effects are rare.

This study will recruit volunteers who continue to have difficult side effects after previous radiotherapy to the pelvis despite receiving the best treatments available from a unique clinic at The Royal Marsden which has pioneered treatment for bowel problems after radiotherapy. Two out of every three volunteers who take part, will be randomly assigned to treatment with Pentoxifylline and Tocovid SupraBio, while one out of three will receive dummy pills. Neither the patients nor the staff assessing them will know which treatment they have been given. Volunteers take the active treatments or dummy tablets for a year and will be assessed regularly while on treatment and for a year afterwards. This study will show whether active treatment is more effective than dummy pills in improving the symptoms caused by radiation-induced fibrosis.

ELIGIBILITY:
Inclusion Criteria -

* Age over 18 years.
* Past history of a malignant pelvic neoplasm (T1-4 N0-2 M0) of the rectum, prostate, testis, bladder, uterine cervix, uterus, vagina, vulva, anal canal or ovary.
* A minimum 12 months follow-up post-radiotherapy (24 months for patients with past history of stage T4 and/or N2 disease).
* A maximum 7 years post-radiotherapy
* No evidence of cancer recurrence.
* Gastrointestinal symptoms attributable to prior radiotherapy: grade 2 or higher in any CTCAE Version 4 category, or grade 1 with difficult intermittent symptoms.
* Symptoms are not relieved by appropriate life-style advice and medication over a 3-month period.
* Physical and psychological fitness for Tocovid SupraBio+PTX therapy.
* Written informed consent and availability for follow up.
* Willingness to keep to a specified level of dietary fat intake during the study.

Exclusion Criteria -

* Surgery for rectal cancer.
* Contra-indication or other inability to undergo magnetic resonance imaging, if required to rule out malignancy.
* Dietary supplementation containing alpha-tocopherol above a daily dose of 30mg at any time during the last three months.
* Medication with pentoxifylline at any time since radiotherapy.
* Pregnancy or breast feeding.
* Ischaemic heart disease, uncontrolled hypertension, hypotension, acute myocardial infarction, cerebral haemorrhage, retinal haemorrhage, renal failure, liver failure and medication with insulin, ketorolac or vitamin K.
* Allergy to soya.
* Known hypersensitivity to the active constituent, pentoxifylline other methyl xanthines or any of the excipients', as per SmPC for pentoxifylline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Change at 12 months in the bowel disease subset of the Modified IBDQ Quality of Life questionnaire. | Endpoint will be assessed pre-treatment and 3, 6, 9, 12, 18 & 24 months post-treatment.

SECONDARY OUTCOMES:
Change at 12 months in rectal IBDQ bleeding score between the two groups in those patients presenting with grade 2, 3 or 4 bleeding. | Endpoint will be assessed pre-treatment and 3, 6, 9, 12, 18 & 24 months post-treatment.
Change at 12 months in IBDQ faecal incontinence score between the two groups in those patients presenting with grade 1 or greater incontinence. | Endpoint will be assessed pre-treatment and 3, 6, 9, 12, 18 & 24 months post-treatment.
Proportion of items graded as marked or severe (grade 3 or 4). | Endpoint will be assessed pre-treatment and 3, 6, 9, 12, 18 & 24 months post-treatment.
Physician assessment of rectal dysfunction based on the modified CTCAE Version 4 grading. | Endpoint will be assessed pre-treatment and 6, 12 & 24 months post-treatment.
Patient self-assessments: QLQ-C30 and CR29 and the Gastrointestinal Symptom Rating Scale. | Endpoint will be assessed pre-treatment and 3, 6, 9, 12, 18 & 24 months post-treatment.
Photographic assessment of rectal mucosa. | Endpoint will be assessed pre-treatment and 12 & 24 months post-treatment
Serum fibrosis marker levels. | Endpoint will be assessed pre-treatment and 3, 6, 9, 12, 18 & 24 months post-treatment.

OTHER OUTCOMES:
Translational endpoint: Rectal biopsies (optional) | Endpoint will be assessed pre-treatment and 12 & 24 months post-treatment.
  Tissue samples will be banked until after the final analysis of the trial, when funding will be sought to identify molecular and cellular correlates of therapeutic response in the event of a statistically significant benefit for Tocovid SupraBio/ PTX combination.
Translational endpoint: Blood samples | Endpoint will be assessed pre-treatment and 12 & 24 months post-treatment.
  Development of novel markers of fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Taylor, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Andreyev HJN, Matthews J, Adams C, Gothard L, Lucy C, Tovey H, Boyle S, Anbalagan S, Musallam A, Yarnold J, Abraham D, Bliss J, Abdi BA, Taylor A, Hauer-Jensen M. Randomised single centre double-blind placebo controlled phase II trial of Tocovid SupraBio in combination with pentoxifylline in patients suffering long-term gastrointestinal adverse effects of radiotherapy for pelvic cancer: The PPALM study. Radiother Oncol. 2022 Mar;168:130-137. doi: 10.1016/j.radonc.2022.01.024. Epub 2022 Jan 29. PMID 35093409